CLINICAL TRIAL: NCT03824808
Title: A Prospective, Randomized, Double-Blinded, Placebo-Controlled Clinical Trial Evaluating the Use of Perioperative Intravenous Lidocaine Infusion to Decrease Pain Scores and Opioid Consumption After Robotic-Assisted Prostatectomy and Robotic-Assisted Partial Nephrectomy
Brief Title: Effect of Perioperative Intravenous Lidocaine Infusion in Robotic-Assisted Urologic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Challenges with recruitment of surgical research subjects in the target population.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Boris Mraovic, Professor of Clinical Anesthesiology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012402
Record Dates: First submitted 2018-11-13; First posted 2019-01-31 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Kidney Cancer; Prostate Cancer
Keywords: prostatectomy; partial nephrectomy; robotic surgery; intravenous lidocaine; lidocaine hydrochloride
MeSH Terms: conditions — Kidney Neoplasms; Prostatic Neoplasms | interventions — Lidocaine; Glucose; Solutions; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will receive either intraoperative 0.8% lidocaine or normal saline at 1 mg/kg/h when younger than 65 years and 0.5 mg/kg/h when greater than or equal to the age of 65 to be delivered by continuous infusion for 24 hours.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeon, anesthesiologist, operating room staff, participant, personnel in the postanesthesia care unit (PACU) as well as the investigators collecting the postoperative data will be blinded to the group allocation. Study medication is prepared and masked by an unblinded investigation drug pharmacist who is not involved in clinical care.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Lidocaine Hydrochloride 0.8% in Dextrose 5% Solution
  Interventions: Drug: Lidocaine Hydrochloride 0.8% in Dextrose 5% Solution
- Control group (Placebo Comparator): 0.9% Sodium Chloride Injection
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Lidocaine Hydrochloride 0.8% in Dextrose 5% Solution — Lidocaine Hydrochloride and 5% Dextrose Injection, USP is a sterile, nonpyrogenic solution prepared from lidocaine hydrochloride and dextrose in water for injection.
  Other Names: Lidocaine
  Arms: Treatment group
Drug: 0.9% Sodium Chloride Injection — Sodium Chloride Injection USP is sterile, nonpyrogenic, isotonic and contains no bacteriostatic or antimicrobial agents.
  Other Names: Normal Saline
  Arms: Control group

SUMMARY:
Controlling pain is fundamental during and after surgical procedures. This study examines pain associated with robotic assisted surgery on prostate cancer or a kidney mass. In recent years, the risk of opioids in the postoperative period has gained interest due to the growing epidemic of addiction, dependence, and overdose. In this study, the investigators expect a continuous infusion of intravenous lidocaine during the perioperative period to result in less pain and less opioid use.

DETAILED DESCRIPTION:
In recent years, the risk of opioids in the post-operative period has gained interest due to the growing epidemic of addiction, dependence, and overdose. The rate of drug overdose secondary to opioids has continued to increase at an alarming rate. This has been a primary point of concern in all fields of medicine and Urology has not been an exception. This is also a nationwide government and public health concern. This has generated an increased focus on the use of non-opioid analgesics after surgery such as intravenous lidocaine.

Opioids remain the primary source of relief for postoperative pain and have the potential to lead to significant morbidity. Opioids may delay recovery following surgery and have many well-known adverse effects including, but not limited to, nausea, vomiting and prolonged post-operative ileus. Furthermore, in one study, they inadequately provided pain control in 50-60% of postoperative participants. This is a frequent report of participants because of the less than optimal utilization of the medications in fear of their dose dependent adverse effects and various contraindications. On the other hand, surplus medication following surgery is another prominent component of the opioid problem in Urologic practices. Bates et al. found that of the 586 participants that underwent a urological procedure that they reviewed, 67% of them had collected surplus medication. It is both necessary and beneficial for surgeons and participants to utilize dose-sparing strategies following surgery to decrease overall opioid usage and outpatient requirement.

One mechanism that has already been employed for overall improvement in prostatectomies and partial nephrectomies is the use of the robotic assisted approach. Robot assisted partial nephrectomies (RALPN) and robotic assisted laparoscopic prostatectomies (RALP) are becoming a mainstay in urologic surgery and increasing annually. This coincides with a continuous downward trend of laparoscopic and open urologic procedures. RALPN has been shown in a meta-analysis to be more favorable than laparoscopic partial nephrectomies and will continue to be the surgical procedure of choice in the near future. RALP is also now the dominant surgical approach while open and laparoscopic prostatectomies becoming less frequent. Robotic assisted surgery is associated with improved functional outcomes, pain scores, shorter hospital stays, and increases in participants satisfaction in many studies.

While there has been a pronounced increase in robotic surgery over the past 10 years that has demonstrated benefits for participants, there has been limited studies regarding the pain management for these participants. Robotic assisted surgery itself decreases pain levels compared to other approaches, but participants continue to experience mild to moderate pain levels in the postoperative period, which are classically managed with NSAIDs and opioids.

Recently, Enhanced Recovery after Surgery protocols (ERAS) have been implemented in an attempt to decrease pain and opioid use as one outcome. ERAS utilizes multimodal analgesia and has shown improvement of participant satisfaction and perioperative opioid use. Systemic lidocaine is becoming more popular and regularly applied through this protocol and, other practices, in due to its analgesic, anti-hyperalgesia and anti-inflammatory properties that it contains. Systemic lidocaine mechanism of action is not fully understood, but it appears to be multifaceted. Systemic lidocaine inhibits voltage-gated sodium channels in both the peripheral and central nervous system. This is believed to cause an additive effect when combined with inhaled anesthetics which also work on the voltage-gated sodium channels in the central nervous system. Despite this summative effect, this is likely not the primary mechanism of action. Instead, it is believed to predominantly act on anti-inflammatory signaling and through inhibiting neuronal effects. Additionally, it reduces nociception and cardiovascular response to surgical stress and pain.

This is a prospective, randomized, double-blinded, placebo-controlled clinical trial on lidocaine infusion for pain control and opioid consumption in participants undergoing either robotic-assisted laparoscopic prostatectomy or robotic-assisted laparoscopic partial nephrectomy at University of Missouri Hospital. Participants will be randomized in a 1:1 fashion and stratified by the type of surgery to receive a perioperative intravenous 0.8% lidocaine infusion at 1 mg/kg/h if < age 65 and 0.5 mg/kg/h if ≥ age 65 or an equal volume and rate of normal saline as a placebo. The infusion will be started 15 minutes after endotracheal intubation and continue for 24 hours.

The study that the investigators propose targets an area of urology that is underrepresented in the current literature despite its increasing importance. To the best of the investigator's knowledge, this has not been directly studied before, although it has been utilized numerous times in the ERAS protocol at the University of Missouri Hospital throughout the Division of Urology and Anesthesiology & Perioperative Medicine in participants undergoing robotic surgery. The benefits of intravenous lidocaine have been demonstrated in other areas and these results warrant a prospective, randomized, double-blinded, placebo controlled study to assess the lidocaine infusion effects for robot assisted laparoscopic prostatectomies and partial nephrectomies. As the number of robotic assisted surgeries and emphasis on opioid reduction continues, the evaluation of systemic lidocaine will be important in improving outcomes in urology.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing robotic assisted prostatectomy or robotic assisted partial nephrectomy at University of Missouri Hospital for prostate cancer or kidney mass
* Age ≥ 18 years
* ASA I-III

Exclusion Criteria:

* Inability to obtain written informed consent
* Allergy to lidocaine or other amide local anesthetics
* Atrioventricular conduction blocks
* CV instability and concomitant use of alpha agonists or beta blockers
* Recent myocardial infarction (≤ 6 months ago)
* Cardiac arrhythmia disorders
* Stokes-Adams syndrome
* Wolff-Parkinson-White syndrome
* Seizure disorders
* Liver failure or hepatic dysfunction
* Significant renal disease with a serum creatinine ≥ 2 mg/dl
* A family history of malignant hyperthermia
* Current use of opioids or documented history of opioid abuse
* Typically, have less than 3 bowel movement per week
* Combined surgical cases that include robotic prostatectomy or robotic partial nephrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Mraovic, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bates C, Laciak R, Southwick A, Bishoff J. Overprescription of postoperative narcotics: a look at postoperative pain medication delivery, consumption and disposal in urological practice. J Urol. 2011 Feb;185(2):551-5. doi: 10.1016/j.juro.2010.09.088. Epub 2010 Dec 18. PMID 21168869
- [Background] Hedegaard H, Warner M, Minino AM. Drug Overdose Deaths in the United States, 1999-2016. NCHS Data Brief. 2017 Dec;(294):1-8. PMID 29319475
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: overdoses of prescription opioid pain relievers---United States, 1999--2008. MMWR Morb Mortal Wkly Rep. 2011 Nov 4;60(43):1487-92. PMID 22048730
- [Background] Dunn LK, Durieux ME. Perioperative Use of Intravenous Lidocaine. Anesthesiology. 2017 Apr;126(4):729-737. doi: 10.1097/ALN.0000000000001527. No abstract available. PMID 28114177
- [Background] De Oliveira GS Jr, Fitzgerald P, Streicher LF, Marcus RJ, McCarthy RJ. Systemic lidocaine to improve postoperative quality of recovery after ambulatory laparoscopic surgery. Anesth Analg. 2012 Aug;115(2):262-7. doi: 10.1213/ANE.0b013e318257a380. Epub 2012 May 14. PMID 22584558
- [Background] Joshi GP, Jaschinski T, Bonnet F, Kehlet H; PROSPECT collaboration. Optimal pain management for radical prostatectomy surgery: what is the evidence? BMC Anesthesiol. 2015 Nov 4;15:159. doi: 10.1186/s12871-015-0137-2. PMID 26530113
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Marcus HJ, Hughes-Hallett A, Payne CJ, Cundy TP, Nandi D, Yang GZ, Darzi A. Trends in the diffusion of robotic surgery: A retrospective observational study. Int J Med Robot. 2017 Dec;13(4):e1870. doi: 10.1002/rcs.1870. Epub 2017 Nov 6. PMID 29105982
- [Background] Choi JE, You JH, Kim DK, Rha KH, Lee SH. Comparison of perioperative outcomes between robotic and laparoscopic partial nephrectomy: a systematic review and meta-analysis. Eur Urol. 2015 May;67(5):891-901. doi: 10.1016/j.eururo.2014.12.028. Epub 2015 Jan 6. PMID 25572825
- [Background] Avulova S, Smith JA Jr. Is Comparison of Robotic to Open Radical Prostatectomy Still Relevant? Eur Urol. 2018 May;73(5):672-673. doi: 10.1016/j.eururo.2018.01.011. Epub 2018 Feb 3. No abstract available. PMID 29398264
- [Background] D'Alonzo RC, Gan TJ, Moul JW, Albala DM, Polascik TJ, Robertson CN, Sun L, Dahm P, Habib AS. A retrospective comparison of anesthetic management of robot-assisted laparoscopic radical prostatectomy versus radical retropubic prostatectomy. J Clin Anesth. 2009 Aug;21(5):322-8. doi: 10.1016/j.jclinane.2008.09.005. Epub 2009 Aug 22. PMID 19700296
- [Background] Batley SE, Prasad V, Vasdev N, Mohan-S G. Post-Operative Pain Management in Patients Undergoing Robotic Urological Surgery. Curr Urol. 2016 Feb;9(1):5-11. doi: 10.1159/000442843. Epub 2016 Feb 10. PMID 26989364
- [Background] Woldu SL, Weinberg AC, Bergman A, Shapiro EY, Korets R, Motamedinia P, Badani KK. Pain and analgesic use after robot-assisted radical prostatectomy. J Endourol. 2014 May;28(5):544-8. doi: 10.1089/end.2013.0783. Epub 2014 Jan 30. PMID 24400824
- [Background] Jendoubi A, Naceur IB, Bouzouita A, Trifa M, Ghedira S, Chebil M, Houissa M. A comparison between intravenous lidocaine and ketamine on acute and chronic pain after open nephrectomy: A prospective, double-blind, randomized, placebo-controlled study. Saudi J Anaesth. 2017 Apr-Jun;11(2):177-184. doi: 10.4103/1658-354X.203027. PMID 28442956
- [Background] Naik BI, Tsang S, Knisely A, Yerra S, Durieux ME. Retrospective case-control non-inferiority analysis of intravenous lidocaine in a colorectal surgery enhanced recovery program. BMC Anesthesiol. 2017 Jan 31;17(1):16. doi: 10.1186/s12871-017-0306-6. PMID 28143397
- [Background] Nakhli MS, Kahloul M, Guizani T, Zedini C, Chaouch A, Naija W. Intravenous lidocaine as adjuvant to general anesthesia in renal surgery. Libyan J Med. 2018 Dec;13(1):1433418. doi: 10.1080/19932820.2018.1433418. PMID 29433385

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Lidocaine Hydrochloride infusion
  The treatment group received a perioperative and intraoperative infusion of 0.8% lidocaine at 1mg/kg/h.
- Control Group: Normal saline
  The control group received normal saline.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 11 patients were randomized into the treatment group, while 10 patients were randomized to the control group. Investigators were blinded to the randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 7 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference in Post-operative Pain Scores Measured by Visual Analog Scale
Description: 10-cm Visual Analog Scale (VAS), score of 0 "no pain" to a score of 10 "worst pain ever"
Time Frame: Through study completion, assessed at 1h, 2h, 4h, 6h, 12h and 24h post operatively, then every 24 hours until discharge, and at the post operative visit which occurred within 21-days post-operatively.
Population: Patients were discharged at different times post operatively, dependent on the procedure performed and post operative pain management. Some patients were discharged before 24 hours post operatively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 11 | 10
score on a scale
  Pain 1 hour post operative | 5.5 (2.8) | 4.0 (2.4)
  Pain 2 hours post operative | 4.4 (3.4) | 4.2 (1.5)
  Pain 4 hours post operative | 4.8 (3.2) | 3.1 (2.2)
  Pain 6 hours post operative | 4.0 (2.1) | 2.5 (2.0)
  Pain 12 hours post operative | 3.6 (2.8) | 2.4 (1.6)
  Pain 24 hours post operative: number analyzed (Participants) | 10 | 8
  Pain 24 hours post operative | 2.3 (1.7) | 1.9 (1.9)
  Pain 48 hours post operative: number analyzed (Participants) | 4 | 1
  Pain 48 hours post operative | 2.5 (2.5) | 2 (0)
  Pain 72 hours post operative: number analyzed (Participants) | 1 | 0
  Pain 72 hours post operative | 5 (0) |
  Pain 96 hours post operative: number analyzed (Participants) | 1 | 0
  Pain 96 hours post operative | 6 (0) |
  Pain 120 hours post operative: number analyzed (Participants) | 1 | 0
  Pain 120 hours post operative | 5 (0) |
  Pain on discharge: number analyzed (Participants) | 3 | 4
  Pain on discharge | 1 (1) | 2 (0)
  Pain at post operative visit: number analyzed (Participants) | 7 | 6
  Pain at post operative visit | 0.5 (1.2) | 0.5 (0.8)

2. Secondary Outcome: Opioid Consumption
Description: Difference in opioid consumption in first 24 hours, discharge and 21 days post-operatively (morphine equivalents)
Time Frame: Through study completion, assessed for first 24-hours post operatively, then every 24 hours until discharge, and at the post operative visit which occurred within 21-days post-operatively.
Population: The milligram morphine equivalent for oral opioid use is reported per group for 24h postop, 25-48h postop, 49-72h postop, 73-96h postop, and 97-120h postop.
Measure: Mean (Standard Deviation); unit: Milligram Morphine Equivalent
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 11 | 10
Milligram Morphine Equivalent
  Milligram morphine equivalent (MME) 0-24h postop: number analyzed (Participants) | 7 | 5
  Milligram morphine equivalent (MME) 0-24h postop | 22.5 (19.4) | 12.0 (5.4)
  Milligram morphine equivalent (MME) 25-48h postop: number analyzed (Participants) | 4 | 2
  Milligram morphine equivalent (MME) 25-48h postop | 26.3 (19.8) | 21.3 (1.8)
  Milligram morphine equivalent (MME) 49-72h postop: number analyzed (Participants) | 1 | 0
  Milligram morphine equivalent (MME) 49-72h postop | 7.5 (0) |
  Milligram morphine equivalent (MME) 73-96h postop: number analyzed (Participants) | 1 | 0
  Milligram morphine equivalent (MME) 73-96h postop | 7.5 (0) |
  Milligram morphine equivalent (MME) 97-120h postop: number analyzed (Participants) | 1 | 0
  Milligram morphine equivalent (MME) 97-120h postop | 7.5 (0) |
  Milligram morphine equivalent (MME) prescribed at discharge for home use | 26.8 (13.8) | 23.0 (7.5)
  Milligram morphine equivalent (MME) used of discharge prescription: number analyzed (Participants) | 5 | 6
  Milligram morphine equivalent (MME) used of discharge prescription | 20.0 (22.6) | 8.8 (12.0)

3. Secondary Outcome: Length of Hospital Stay
Description: Difference in length of hospital stay determined by surgeon excluding social factors that may delay discharge
Time Frame: At participant discharge, assessed up to 14 days (+/-) 7 days
Population: Patients were discharged at different times, dependent on post operative recovery and pain management.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 11 | 10
Participants
  Discharged within 24 hours | 1 | 2
  Discharged between 24 and 48 hours | 6 | 7
  Discharged between 48 and 72 hours | 3 | 1
  Discharged between 72 and 96 hours | 0 | 0
  Discharged between 96 and 120 hours | 0 | 0
  Discharged between 120 and 144 hours | 1 | 0

4. Secondary Outcome: Duration of Post-operative Ileus
Description: Difference in post-operative Ileus duration
Time Frame: as for outcome 1
Population: Patients were discharged mostly within 48 hours post operatively, and post operative follow up was not successful. This is not a reliable result.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 11 | 10
Participants
  Total patients recorded with returned ileus at 1 hour postop | 0 | 0
  Total patients recorded with returned ileus at 2 hours postop | 0 | 0
  Total patients recorded with returned ileus at 4 hours postop | 0 | 0
  Total patients recorded with returned ileus at 6 hours postop | 0 | 0
  Total patients recorded with returned ileus at 12 hours postop | 0 | 0
  Total patients recorded with returned ileus at 24 hours postop | 0 | 1
  Total patients recorded with returned ileus at 48h postop | 1 | 0
  Total patients recorded with returned ileus at 72 hours postop | 1 | 0
  Total patients recorded with returned ileus at 96 hours postop | 0 | 0
  Total patients recorded with returned ileus at 120 hours postop | 0 | 0
  Total patients who did not have returned ileus on discharge | 9 | 9

5. Secondary Outcome: Post-operative PACU Time
Description: Difference in time in the Post Anesthesia Care Unit (PACU) after surgery
Time Frame: During hospitalization, approximately 2 hours post-surgery
Population: Data were not captured for 9 patients in the treatment group and 8 patients in the control group.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 2 | 2
Minutes | 59 (7.8) | 122.5 (53)

6. Secondary Outcome: Return of Flatus
Description: Difference in return of flatus after surgery
Time Frame: During hospitalization at 1h, 2h, 4h, 6h, 12h, and 24h post operatively, then every 24 hours thereafter until discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 11 | 10
Participants
  Return of flatus 2 hours post operative | 0 | 1
  Return of flatus 4 hours post operative | 1 | 0
  Return of flatus 6 hours post operative | 1 | 2
  Return of flatus 12 hours post operative | 5 | 2
  Return of flatus 24 hours post operative | 4 | 5

7. Secondary Outcome: Time to Out of Bed
Description: Difference in time to out of bed to chair after surgery
Time Frame: During hospitalization regular intervals for the first 24 hours, then every 24 hours until discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 11 | 10
Participants
  Out of bed to chair 2 hours post operative | 0 | 1
  Out of bed to chair 4 hours post operative | 0 | 0
  Out of bed to chair 6 hours post operative | 1 | 1
  Out of bed to chair 12 hours post operative | 2 | 1
  Out of bed to chair 24 hours post operative | 3 | 5
  Out of bed to chair 48 hours post operative | 2 | 0
  Patients out of bed to chair only at discharge | 0 | 1
  Patients not recorded | 3 | 1

8. Secondary Outcome: First Ambulation in the Hallway
Description: Difference in time to first ambulation in the hallway after surgery
Time Frame: During hospitalization at 1h, 2h, 4h, 6h, 12h, and 24h post operatively, then every 24 hours until discharge.
Population: Number of patients ambulated at 1h, 2h, 4h, 6h, 12h, 24h post-operatively, then recorded every 24h until discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 11 | 10
Participants
  Ambulated 6 hours post operatively | 1 | 0
  Ambulated 12 hours post operatively | 3 | 1
  Ambulated 24 hours post operatively | 3 | 6
  Ambulated 48 hours post operatively | 0 | 0
  Ambulated 72 hours post operatively | 0 | 0
  Patients who only ambulated at discharge | 0 | 1
  Patients who did not ambulate by discharge | 2 | 2
  Patients not recorded | 2 | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored during hospitalization until the postoperative visit which occurred within 21 days after discharge.
Description: The study followed the ClinicalTrials.gov definitions of adverse/serious adverse events for collection of information.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT03824808/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT03824808/ICF_004.pdf